CLINICAL TRIAL: NCT03281616
Title: Lifestyle Interventions in Turkish-background Patients With Metabolic Syndrome and Diabetes in Germany
Brief Title: Lifestyle in Turkish-Background Diabetics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Michael Boschmann, Physician, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Refine
Record Dates: First submitted 2017-09-11; First posted 2017-09-13 (Actual); Last update posted 2017-09-19 (Actual); Status verified 2017-09

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus | interventions — Diet

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diet and Physical Activity Recording (Active Comparator)
  Interventions: Behavioral: Diet
- Diet and No Physical Activity Recording (Active Comparator)
  Interventions: Behavioral: Diet

INTERVENTIONS:
Behavioral: Diet — Individually tailored diets; 30% caloric reduction according to daily energy requirements measured by indirect calorimetry

SUMMARY:
Background: Life-style interventions are indicated in patients with metabolic syndrome and/or type 2 diabetes. However, cultural differences are substantial confounders to not only compliance, but also whether or not the interventions are offered in the first place. In Germany, the large Turkish-background minority has a particularly high incidence of type 2 diabetes, but there is no recorded evidence of a life-style intervention in this patient group.

Objective: The investigators tested the body weight-reducing effect of a 30% calorie-reduced diet, adjusted to individual eating habits and preferences regarding quality and resources of food in a Turkish-background cohort.

DETAILED DESCRIPTION:
The investigators conducted a prospective, randomized, two-arm parallel study. In both arms, patients were instructed in a 12-week diet that was reduced by in caloric content by at least 30% based on calorimetric measurements of 24 h resting energy expenditure and estimated additional expenditures by diet- and activity-induced thermogenesis. Before and after the diet, anthropometric measures and various MetS-associated blood parameters were determined.

The subjects were not instructed in an exercise program. However, the subjects were advised on the value of increased physical activity. For additional motivation, effects were tested by an activity monitor. Therefore, in one of the arms, 24 hour locomotor activity and energy expenditure were determined by means of the SenseWear® MF armband (Body Media Inc., AliphCom dba Jawbone®, Pittsburgh, PA, U.S.A.). This device detects activity contest using accelerometers and assesses daily energy expenditure. For allocation of the subjects, a computer-generated list of random numbers was used. The randomization sequence was created using SPSS 18 (SPSS, Inc., Chicago, IL, USA) statistical software and subjects were assigned to be tested or not for locomotor activity with a 1:1 allocation using random block sizes of 2, 4, and 6.

ELIGIBILITY:
Inclusion Criteria:

* Age 30 - 65 years
* BMI 30 - 40 kg/m2
* non-Insulin dependent diabetes

Exclusion Criteria:

* Pregnancy
* more than 3 anti-diabetic drugs

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2014-06-01 (Actual); Primary Completion 2015-06-30 (Actual); Study Completion 2015-09-30 (Actual)

PRIMARY OUTCOMES:
Body weight reduction | 12 weeks
  Changes in body weight (kg) within 12 weeks of diet

SECONDARY OUTCOMES:
Blood glucose | 12 weeks
  Changes in blood glucose (mmol/L) within 12 weeks of diet
Blood HbA1c | 12 weeks
  Changes in blood glycated hemoglobin within 12 weeks of diet

IPD SHARING:
Plan to Share IPD: No